CLINICAL TRIAL: NCT03713671
Title: The Effect of Quadriceps Femoris Muscle Fatigue Protocol on Gait and Balance Parameters Before and After Parathyroidectomy in Patients With Primary Hyperparathyroidism
Brief Title: Gait and Balance Parameters Before and After Parathyroidectomy in Patients With Primary Hyperparathyroidism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Recep Tayyip Erdogan University Training and Research Hospital (Other)
Collaborators: Hacettepe University (Other); Ankara Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Melek Merve ERDEM, Research Assistant, Recep Tayyip Erdogan University Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: GO 18/790
Record Dates: First submitted 2018-10-18; First posted 2018-10-22 (Actual); Last update posted 2023-12-05 (Actual); Status verified 2023-12

CONDITIONS: Primary Hyperparathyroidism
Keywords: Primary Hyperparathyroidism; Spatio-Temporal Parameters of Gait; Gait Symmetry; Balance
MeSH Terms: conditions — Hyperparathyroidism, Primary | interventions — Gait Analysis

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PHPT Group (Other): Spatio-Temporal gait analysis and balance assessment of subjects with Primary Hyperparathyroidism
  Interventions: Diagnostic Test: gait analysis
- Control Group (Other): Spatio-Temporal gait analysis and balance assessment of healthy subjects
  Interventions: Diagnostic Test: gait analysis

INTERVENTIONS:
Diagnostic Test: gait analysis — Computerized gait analysis system will use to evaluate spatio-temporal gait parameters

SUMMARY:
This study will evaluate how Quadriceps Femoris muscle fatigue protocol affect the spatio-temporal gait parameters, gait symmetry and balance in individuals with primary hyperparathyroidism before and after parathyroidectomy. Study group will consist of 20 subjects with primary hyperparathyroidism (PHPT) and control group will consist of 20 healthy subjects.

DETAILED DESCRIPTION:
Parathyroid hormone, released from the parathyroid gland, plays an important role in keeping the ionized calcium in between the reference values in body. Precise control of ionized calcium is particularly necessary to ensure the optimal function of physiological processes such as providing intracellular signaling, performing neuromuscular functions and bone metabolism. When there is a decrease in the level of ionized calcium in the systemic circulation due to any reason, increased calcium concentration is maintained as a result of the increased absorption of calcium from the kidneys, bones and intestines into the blood via increased parathyroid hormone. An error caused by any of the components in this regulatory system may cause excessive parathyroid hormone release, causing primary, secondary or tertiary hyperparathyroidism. Primary hyperparathyroidism (PHPT) is a common endocrinological disorder, which is characterized by excessive release of parathyroid hormone, resulting in a defect in the regulation of calcium metabolism. PHPT, is the third most common endocrine disease and is the most common cause of hypercalcemia. Today, PHPT is approximately 0.25-0.66% of the population and it is seen as 3: 1 times more common in women than men. While the incidence of the disease increases with age, it increases dramatically after 50 years of age. The clinical presentation of PHPT ranges from asymptomatic disease to the classical symptomatic disease of renal and / or musculoskeletal complications. Low plasma 25 Hydroxyvitamin D level; bone mineral density, muscle strength, preservation of postural stability and functional performance of the musculoskeletal functions such as disruption caused by the person's walking and balance activities are adversely affected.In addition, fatigue, pain, and body mass index, as a result of the increase in the functional capacity of the person is seriously reduced quality of life and psychosocial status is adversely affected. Although there are studies related to bone mineral density, muscle strength and function, instability, fatigue, etc., which are secondary to PHPT and cause a significant decrease in functional capacity, there is no study to investigate the effect of M. quadriceps Femoris ,which has a key role in the evaluation of functional capacity, muscle fatigue on the gait and balance parameters in the pre and post-treatment period in the literature. The aim of this case-control study is to investigate the effect of Quadriceps Femoris muscle fatigue protocol on gait, gait symmetry and balance parameters before and after parathyroidectomy in patients PHPT and to compare that parameters of these individuals with healthy controls with similar demographic characteristics that included in the control group.

ELIGIBILITY:
Inclusion Criteria:

* PHPT group, include cases with a Primary Hyperparathyroidism
* Control group consists of healthy adults with the similar demographic characteristics as study group.

Exclusion Criteria:

* The presence of osteoarticular deformities
* Walking with assist device
* Having a neurological disease that may affect the performance
* To have significant and irreversible visual deficits
* The body mass index (BMI) is greater than> 40 kg / m²
* There is an inability to prevent any of the tests
* Individuals with cancer history and chemotherapy (over the last 5 years)
* Plasma creatinine level> 150 µmol / L
* Use of Cinacalcet or Etalpha
* Having a history of diabetes mellitus

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-10-17 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-08-27 (Actual)

PRIMARY OUTCOMES:
Step Length | 1 week
  It is measured along the length of the walkway, from the heel center of the current footprint to the heel center of the previous footprint on the opposite foot.The unit of measure is centimeters.

SECONDARY OUTCOMES:
Stride Length | 1 week
  It is measured on the line of progression between the heel points of two consecutive footprints of the same foot (left to left, right to right). The unit of measure is centimeters.
Static Balance Assessment | 1 week
  The Romberg test will use to assessment for diagnose sensory ataxia, a gait disturbance caused by abnormal proprioception involving information about the location of the joints. The Static Balance Assessment of the individuals in the PHPT group were assessed before and 3 months after Parathyroidectomy.
Dynamic Balance Assessment | 1 week
  To determine fall risk and measure the progress of balance, sit to stand, and walking Timed Up and Go Test will use. The Dynamic Balance Assessment of the individuals in the PHPT group were assessed before and 3 months after Parathyroidectomy.
Fatigue Severity | 1 week
  The fatigue level that individuals perceived during the performance was recorded using the Fatigue Severity Scale. This is a nine-items questionnaire that assesses the effect of fatigue on daily living. Each item is a statement on fatigue that the subject rates from 1, ' strongly disagree ' to 7, ' strongly agree '.
Functional Capacity | 1 week
  6 Minute Walk test was used to evaluate the functional capacity. The test was performed in a corridor on a flat hard surface of 30 m in length in a straight line. Before the examination, the patient rested for 10 min in a sitting position. It is calculated by measuring the distance that the person walks at the end of this period by asking the person to walk for 6 minutes along a 30 m corridor. In cases of chest pain, dyspnea, leg cramps, excessive fatigue, sweating and wilting, the test should be terminated immediately. The clinician supervising the test instructed the subject on the walking technique and the possibility of taking a rest. At one-minute intervals during the test, the participant received information about the time remaining until the end of the test.
Step Width | 1 week
  It is measured from the midline midpoint of the current footprint to the midline midpoint of the previous footprint on the opposite foot.The unit of measure is centimeters.
Foot Progression Angle | 1 week
  It is the angle between the line of progression and the midline of the footprint. This angle is zero if the geometric mid- line of the footprint is parallel to the line of progression; positive, toe-out, when the mid-line of the footprint is outside the line of progression and negative, toe-in, when inside the line of progression. The unit of measure is degrees.
Speed | 1 week
  It is obtained after dividing the distance traveled by the ambulation time. It is expressed in centimeters per second (cm/sec)
Cadence | 1 week
  The rate at which a person walk, expressed in steps per minute (step/min). The average cadence is 100 - 115 steps/min.
Percentage of Double Support | 1 week
  It is the amount of time that a person spends with both feet on the ground during one gait cycle. It is presented as a percentage of the gait cycle time (% gait cycle). The percentage of time spent in double support decreases as the speed of walking increases.
Percentage of Stance | 1 week
  The stance phase is the weight bearing portion of each gait cycle. It is initiated by heel contact and ends with toe off of the same foot. It is the time elapsed between the first contact and the last contact of two consecutive footfalls on the same foot. It is also presented as a percentage of the gait cycle time (% gait cycle)
Percentage of Swing | 1 week
  It is initiated with toe off and ends with heel strike. It is the time elapsed between the last contact of the current footfall to the first contact of the next footfall on the same foot. It is expressed in seconds (sec) and it is also presented as a percent of the gait cycle (% gait cycle) of the same foot. The Swing Time is equal to the Single Support time of the opposite foot.
Gait Symmetry | 1 week
  It's calculated in order to evaluate symmetry and bilateral coordination of gait. The Symmetry Index and Symmetry Angle are interpreted as a complete symmetry if the result is 0. Evaluation of asymmetries observed in the spatio-temporal characteristics, a deviation of at least 10% from the 0 value for exact symmetry.

CONTACTS AND LOCATIONS:
Overall Officials: Melek M. ERDEM, Principal Investigator — Tayyip Erdogan University Training and Research Hospital; Gonul KOC, MD, Study Director — Ankara Education and Research Hospital; Semra TOPUZ, Assoc. Prof., Study Director — Hacettepe University; Mikail K. DEMIREL, MD, Study Chair — Ankara Education and Research Hospital; Cavit CULHA, Assoc. Prof., Study Chair — Ankara Education and Research Hospital
Locations (1):
- Ankara Education and Research Hospital, Ankara, Cankaya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data for all primary and secondary outcome measures will be made available.
Supporting Information: Study Protocol, CSR
Time Frame: Data will be available within 6 months with completion of the result report.
Access Criteria: Requestors will be required to sign a Data Access Agreement.
URL: https://orcid.org/0000-0003-4073-3084

REFERENCES:
- [Background] Rolighed L, Rejnmark L, Sikjaer T, Heickendorff L, Vestergaard P, Mosekilde L, Christiansen P. No beneficial effects of vitamin D supplementation on muscle function or quality of life in primary hyperparathyroidism: results from a randomized controlled trial. Eur J Endocrinol. 2015 May;172(5):609-17. doi: 10.1530/EJE-14-0940. Epub 2015 Feb 2. PMID 25646406